CLINICAL TRIAL: NCT00504517
Title: Preparing the Personal Physician for Practice (P4)
Acronym: P4
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: 27074
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: Outpatient continuity training; Relevant, Patient-centered curriculum; Evaluation; New graduation requirements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Evaluating Educational Models — Evaluating various forms of educational models for physicians.

SUMMARY:
We would like to better understand how different educational strategies may influence the practice of family medicine. More specifically, we are interested in participant satisfaction with the educational program, participant retainment in this career, and to see if the curricular change better prepares participants for contemporary clinical practice.

DETAILED DESCRIPTION:
In 2004, the Future of Family Medicine report called for implementation of innovative strategies in residency education, allowing translational key insights from the national demonstration project toward new approaches to family medicine training. Taking full advantage of the P4 Project will require careful evaluation planning and implementation. A comprehensive evaluation plan for the P4 Project will be implemented by a core evaluation team that will interact with site-specific evaluators.

The P4 evaluation program represents an observational case series assessment of selected residency programs. It is not an intervention trial; rather each residency program will systematically enroll cohorts of learners who will be exposed to curricular content and learning approaches that will likely be innovative and unique. In the absence of a rigorous study design, core data elements should be obtained from each program including: learner characteristics, program characteristics, and both nationally available data and targeted validated instruments that can link specific educational interventions to learners knowledge, attitudes and skills.

ELIGIBILITY:
Inclusion Criteria:

* Medical Residents at Christiana Care's Residency Program

Ages: 26 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All Family medicine residents who accept employment as a resident in the Dept of Family Medicine will be part of the study population. These residents are interviewed prior to acceptance. Acceptance can occur via the NRMP or osteopathic match process or outside of the match
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa C Maxwell, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health System, Wilmington, Delaware, United States